CLINICAL TRIAL: NCT02815891
Title: A Longitudinal Observational Study of Patients With Nonalcoholic Steatohepatitis (NASH) and Related Conditions Across the Entire Spectrum of Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-NASH
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-NASH will be invited to participate in the Biorepository Specimen Bank (BSB). Blood samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the patient's unique study ID number and the date that the sample was obtained. This link between the patient's study ID number and their name will be available only at the site where the samples were obtained.
Oversight: Data Monitoring Committee: No

SUMMARY:
TARGET-NASH is a longitudinal observational cohort study of patients being managed for NASH and related conditions across the entire spectrum NAFLD in usual clinical practice. TARGET-NASH is a research registry of patients with NAFL or NASH within academic and community real-world practices maintained in order to assess the safety and effectiveness of current and future therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Adults and children (age 2 or older) being managed or treated for nonalcoholic fatty liver disease. Diagnosis is based on the clinical judgement of the care provider.

Exclusion Criteria:

1. Inability to provide informed assent/consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with NAFL or NASH who are being seen specifically to address this disease process
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-07; Primary Completion 2036-07 (Estimated); Study Completion 2036-07 (Estimated)

PRIMARY OUTCOMES:
Establish an understanding of the current natural history of NASH at academic and community medical centers | 10 years
  A detailed analysis of demographics, concurrent medications, metabolic and cardiovascular co-morbidities, staging of liver disease, and outcomes for patients with NASH managed in diverse clinical settings will serve as an important comparator for subsequent interventions that alter the treatment paradigm for this disease.
Evaluate NASH treatment regimens being used in clinical practice | 10 years
  Currently, there are no FDA approved therapies for NASH, however clinicians may use a variety of interventions including diet and exercise programs, vitamin E, bariatric surgery or other unapproved uses of some cholesterol, lipid lowering, anti-diabetic and anti-inflammatory medications as well as alternative medications. TARGET-NASH will monitor the safety and effectiveness of the various treatment choices in enrolled patients.
Examine populations underrepresented in phase II-III clinical trials | 10 years
  Patients with cirrhosis, age > 70, patients who consume moderate amounts of alcohol and patients with multiple comorbidities such as severe depression, chronic fatigue, fibromyalgia, type 2 diabetes, inflammatory bowel disease, or cardiovascular disease.
Evaluate optimal duration and combination of NASH therapies to achieve clinical response and clinical remission | 10 years
  In addition to diet and exercise, type, dose and duration of therapy of each NASH treatment (both current unapproved therapies and future FDA approved drugs) will be closely followed, with a goal to monitor treatment paradigms and various combination regimens for clinical response and clinical remission.
Examine liver histology | 10 years
Estimate adverse event frequency and severity and describe management practices | 10 years
  NASH can often be an asymptomatic disease in the setting of other disease-related comorbidities such as diabetes and cardiovascular disease. Once NASH progresses to cirrhosis, these patients can suffer the attendant complications of decompensated liver disease including debilitating fatigue, muscle wasting, ascites, bleeding, encephalopathy, hepatocellular carcinoma, and death. NASH therapies may increase the frequency and severity of certain adverse events, such as edema (pioglitazone), some cancers (vitamin E), and new agents or combinations of agents may have their own unique adverse event profiles and varying needs for management plans (e.g., pruritus and dyslipidemia).
Evaluate the impact of NASH therapies on medical co-morbidities | 10 years

CONTACTS AND LOCATIONS:
Locations (74):
- United States (67):
  - Banner University Medical Center - Phoenix Transplant Center and Advanced Liver Clinic, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California, Davis, Sacramento, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Connecticut Gastroenterology, Hartford, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Medstar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - Gastro Florida, Clearwater, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - UF Health Gastroenterology, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Schiff Center for Liver Disease/University of Miami, Miami, Florida
  - AdventHealth Diabetes Institute, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Emory University - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Northwestern Medicine, Digestive Health Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Indiana University - Division of Gastroenterology and Hepatology, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Houma Digestive Health Specialists, Houma, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University - Gastroenterology and Hepatology, Clinical Research Unit, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NorthWell Health - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Children's Hospital at Montefiore, Division of Pediatric GI, The Bronx, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Center for Liver Disease and Transplant at CMC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastroenterology Associates, Greenville, South Carolina
  - Children's Health - Children's Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Germany (3):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Aachen, Aachen
  - Charite Berlin, Berlin
- Spain (4):
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Virgen del Rocio, Seville
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanyal AJ, Munoz B, Cusi K, Barritt AS 4th, Muthiah M, Mospan AR, Reddy KR, Firpi-Morell R, Thuluvath PJ, Bhamidimarri KR, Fried MW; TARGET-NASH Investigators. Validation of a Clinical Risk-based Classification System in a Large Nonalcoholic Fatty Liver Disease Real-world Cohort. Clin Gastroenterol Hepatol. 2023 Oct;21(11):2889-2900.e10. doi: 10.1016/j.cgh.2023.02.024. Epub 2023 Mar 5. PMID 36871772
- [Derived] Malespin MH, Barritt AS 4th, Watkins SE, Schoen C, Tincopa MA, Corbin KD, Mospan AR, Munoz B, Trinh HN, Weiss LM, Reddy KR, Loomba R, Kemmer N, Lok AS. Weight Loss and Weight Regain in Usual Clinical Practice: Results From the TARGET-NASH Observational Cohort. Clin Gastroenterol Hepatol. 2022 Oct;20(10):2393-2395.e4. doi: 10.1016/j.cgh.2021.01.023. Epub 2021 Jan 21. PMID 33486083
- [Derived] Weinberg EM, Trinh HN, Firpi RJ, Bhamidimarri KR, Klein S, Durlam J, Watkins S, Reddy KR, Weiss M, Zink RC, Lok AS. Lean Americans With Nonalcoholic Fatty Liver Disease Have Lower Rates of Cirrhosis and Comorbid Diseases. Clin Gastroenterol Hepatol. 2021 May;19(5):996-1008.e6. doi: 10.1016/j.cgh.2020.06.066. Epub 2020 Jul 3. PMID 32629123